CLINICAL TRIAL: NCT02883348
Title: Satisfaction With Care and Quality of Life After Hospital Stay for Chronic Disease
Brief Title: Satisfaction With Care and Quality of Life
Acronym: SATISQOL
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Other Study IDs: Satisqol
Record Dates: First submitted 2016-08-23; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Investigating the predictive value of patient satisfaction with care on 6 months and 1-year quality of life.

DETAILED DESCRIPTION:
Background: Evaluating the impact of complex procedures of patient care for chronic disease patients is one of the objectives and priorities defined in the French framework of the Public Health Act of August 2004. The relevant indicators that predict the impact of the medium-term hospitalization on the quality of life remain to be explored.

Preliminary data showed that care satisfaction, usual indicator of quality of care, was associated with quality of life away from the hospital, especially in the field of orthopedics (prosthetic surgery). Satisfaction is an indicator currently collected in routine periodic surveys in all establishments. This project will test the hypothesis of the prognostic role of this satisfaction after a medical or a surgical treatment in people hospitalized for chronic disease.

Objective: The objective of this research is to investigate the prognostic value of satisfaction with care on the quality of life of patients with chronic disease hospital, at 6 months and 1 year of discharge.

Patients and methods: A multicenter cohort of 1520 patients hospitalized in medical and surgical units for chronic disease (in the field of cardiovascular, musculoskeletal, nephrology, urology, digestive, pulmonary or endocrine). Patients will respond to PJHQ satisfaction questionnaire at the waning of their hospital stay. The quality of life (SF-36) will be measured at 6 months and 1 year after hospitalization.

The socio-demographic characteristics, diagnosis, anxiety state (HAD), optimistic / pessimistic personality (LOT-R), comorbidities (Charlson and Functional comorbidity index), major health events (rehospitalization, death ) and the characteristics of the stays and care structure (cluster services) who welcomed them will be saved.

The number of subjects required was calculated based on a cluster sampling (13 poles or services between institutions) to highlight with a power of 80% a difference of 5 points of quality of life among the satisfied and less satisfied subjects.

Statistical analysis will study the relationship of satisfaction scores with QoL dimensions at 6 months and 1 year, in hierarchical regression multilevel models adjusted for confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-75 years
* Patients hospitalized for treatment of chronic disease, defined as a disease lasting for more than 6 months, and confirmed by a validation committee
* Hospitalization motivation is:

  * A care of an acute episode of a chronic disease
  * A car of a worsening of chronic disease
  * A new therapeutic of a chronic disease

Exclusion Criteria:

* Patients who did not have a therapeutic intervention during their hospitalization (i.e., diagnostic analysis or medical follow-up without change of their treatment)
* Patients with more than 5 hospitalizations during the previous 5 years (more than 1 per year)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population-based
Sampling Method: Probability Sample
Enrollment: 1520 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life score | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Francis GUILLEMIN, MD, PhD, Principal Investigator — CHRU NANCY

IPD SHARING:
Plan to Share IPD: Yes
open to partnership